| Participant No.: | Date: |
|------------------|-------|



## Department of Psychiatry | The University of Hong Kong <u>Consent Form</u>

## The Effectiveness of Repetitive Transcranial Magnetic Stimulation (rTMS) on Improving Sleep Quality in Adults Without Serious Mental Illness

Principal Investigator: Dr. Cheng Pak Wing, Assistant Professor, Department of Psychiatry, Faculty of Medicine, The University of Hong Kong

| 1 | The participant has read and understood to dated//, and have had the opportunity | | for the study |
|---|---|---|---|
| 2 | The participant understands that participal may withdraw at any time without provide affecting our medical care or legal rights. | ing any reason, and v | |
| 3 | The participant understands that in relation Department of Psychiatry of The University of Hong Kong itself, the Institutional Personal Psychiatry | on to this study, person ity of Hong Kong, The Board of the Uniong West Cluster, or redical records. The p | ne University<br>iversity of<br>egulatory |
| 4 | The participant is required to undergo <u>six</u> sessions of repetitive transcranial | | |
| 5 | The participant agrees that the researchers may contact us in the future using the contact details provided in this study for related research purposes. | | |
| 6 | 6 All procedures involved in the study are provided free of charge. | | |
| 7 | There are no conflicts of interest regarding the use of the rTMS machine in this study that influenced the design, implementation, or interpretation of the research. | | |
| Na | ame of the participant D | Date | Signature |
| Na | Vame of the researcher | Pate | Signature |